CLINICAL TRIAL: NCT00383695
Title: A Multicentre Randomised Phase II Clinical Trial Comparing Oxaliplatin (Eloxatin), Capecitabine (Xeloda) and Pre-Operative Radiotherapy With or Without Cetuximab Followed by Total Mesorectal Excision for the Treatment of Patients With Magnetic Resonance Imaging (MRI) Defined High Risk Rectal Cancer
Brief Title: Oxaliplatin, Capecitabine, and Radiation Therapy With or Without Cetuximab in Treating Patients Undergoing Surgery for High-Risk Rectal Cancer
Acronym: EXPERT-C
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000503948; RMNHS-RMH-CCR-2553; EU-20635; EUDRACT-2004-004707-38; CRUK-EXPERT-C; MERCK-RMNHS-RMH-CCR-2553
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the rectum; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Cetuximab; Capecitabine; Oxaliplatin; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: cetuximab
Drug: capecitabine
Drug: oxaliplatin
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving chemotherapy and radiation therapy with or without cetuximab before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. It is not yet known whether giving oxaliplatin, capecitabine, and radiation therapy is more effective with or without cetuximab when given before surgery in treating rectal cancer.

PURPOSE: This randomized phase II trial is studying oxaliplatin, capecitabine, and radiation therapy to compare how well they work with or without cetuximab in treating patients undergoing surgery for high-risk rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the pathological complete response rate at total mesorectal excision in patients with high-risk rectal cancer treated with neoadjuvant therapy comprising oxaliplatin, capecitabine, and radiotherapy with or without cetuximab.

OUTLINE: This is a multicenter, open-label, randomized, controlled study. Patients are stratified according to participating center and presence of T4 disease (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I:

  * Neoadjuvant chemotherapy: Patients receive oxaliplatin IV over 2 hours on days 1, 22, 43, and 64 and oral capecitabine twice daily on days 1-14, 22-35, 43-56, and 64-77.
  * Neoadjuvant chemoradiotherapy: Patients undergo radiotherapy once daily on days 85-89, 92-96, 99-103, 106-110, 113-117, and 120-124 and receive oral capecitabine twice daily on days 85-126.
  * Surgery: Four to six weeks after completion of chemoradiotherapy, patients undergo total mesorectal excision (TME).
  * Adjuvant therapy: Beginning 6-8 weeks after surgery, patients receive oxaliplatin IV over 2 hours on days 1, 22, 43, and 64 and oral capecitabine twice daily on days 1-14, 22-35, 43-56, and 64-77.
* Arm II:

  * Neoadjuvant therapy: Patients receive oxaliplatin and capecitabine as in arm I neoadjuvant chemotherapy and cetuximab IV over 1-2 hours on days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
  * Neoadjuvant chemoradiotherapy: Patients undergo radiotherapy and receive capecitabine as in arm I neoadjuvant chemoradiotherapy and cetuximab IV over 1 hour on days 85, 92, 99, 106, 113, and 120.
  * Surgery: Four to six weeks after completion of chemoradiotherapy patients undergo TME as in arm I.
  * Adjuvant therapy: Beginning 6-8 weeks after surgery, patients receive oxaliplatin and capecitabine as in arm I adjuvant chemotherapy and cetuximab IV over 1 hour on days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed periodically.

After completion of study treatment, patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually for 2 years.

PROJECTED ACCRUAL: A total of 164 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma or undifferentiated non-small cell carcinoma of the rectum
* MRI-defined high-risk, operable disease, defined by ≥ 1 of the following:

  * Tumors within 1 mm of mesorectal fascia (i.e., circumferential resection margin threatened or involved)
  * T3 tumors at or below levators
  * Tumors extending ≥ 5 mm into perirectal fat
  * T4 tumors
  * Presence of extramural venous invasion (primary tumor is therefore at least T3)
* No evidence of metastatic disease by CT scan of the chest and abdomen or, if required, by positron emission tomography scan or biopsy
* No rectal cancer that is unlikely to be operable even after neoadjuvant treatment (i.e., tumor involving the internal iliac vessels)
* No T1-2 rectal cancer, in the absence of other high-risk factors

  * T2 tumors within 1 mm of mesorectal fascia allowed
* No recurrent disease

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy > 3 months
* WBC > 3,000/mm³
* Absolute neutrophil count > 1,500/mm³
* Platelet count > 100,000/mm³
* Bilirubin < 1.5 times upper limit of normal (ULN)
* Transaminases < 2.5 times ULN
* Creatinine normal OR creatinine clearance > 50 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No concurrent uncontrolled medical condition
* No other active malignant disease within the past 10 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No contraindications to MRI (e.g., pacemaker)
* No medical or psychiatric conditions that would preclude informed consent
* No known malabsorption syndrome or lack of physical integrity of the upper gastrointestinal tract
* No clinically significant (i.e., active) cardiac disease, including any of the following:

  * Congestive heart failure
  * Symptomatic coronary artery disease
  * Cardiac dysrhythmia (e.g., atrial fibrillation, even if controlled with medication)
  * Myocardial infarction within the past 12 months
* No symptoms or history of peripheral neuropathy

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy, radiotherapy, or investigational treatment for rectal cancer
* No other concurrent cytotoxic agents or investigational drugs
* No concurrent sorivudine or sorivudine analogues (e.g., brivudine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2005-09

PRIMARY OUTCOMES:
Pathological complete response rate at time of total mesorectal excision (TME)

SECONDARY OUTCOMES:
Radiological response rates after completion of neoadjuvant therapy
Complete resection rate (R0 resection) with microscopic clear resection margin (tumor observed > 1 mm from the resection margin), especially circumferential resection margin
Perioperative measures, including operation time, duration of in-patient stay, perioperative transfusion requirement, and mortality, within 30 days of TME
Postoperative complications, including wound infection, wound dehiscence, and fistula formation
Quality of TME as assessed by audit of photographed surgical specimens
Rate of abdominoperitoneal excision
Rate of permanent defunctioning colostomies
Clinical and radiological anastomotic leak rate
Progression-free survival and patterns of failure
Overall survival
Safety
Quality of life, including long-term bowel function

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, MD, Study Chair — Royal Marsden NHS Foundation Trust
Locations (13):
- Spain (3):
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- Sweden (2):
  - Karolinska University Hospital - Solna, Stockholm
  - Uppsala University Hospital, Uppsala
- United Kingdom (8):
  - Royal Bournemouth Hospital NHS Trust, Bournemouth, England
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Eastbourne District General Hospital, Eastbourne, England
  - Cancer Research UK Clinical Groups at Guy's King's & St. Thomas' Hospitals, London, England
  - Mid Kent Oncology Centre at Maidstone Hospital, Maidstone, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England